CLINICAL TRIAL: NCT05808868
Title: Identify Patients at Risk of Moderate or Severe OSA During ENT Examination
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Duc Trung Nguyen, MD, PhD, Dr NGUYEN Duc Trung - Hospital practitioner, Central Hospital, Nancy, France
Other Study IDs: 2021PI120
Record Dates: First submitted 2023-03-25; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Sleep Apnea Syndromes
Keywords: SAOS
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSA screening: To
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — The detailed management is not different from that usually practiced in our department.
  Each patient benefits from an ENT consultation where an interrogation is carried out concerning the sleep disorders, the answer to the usual questionnaires screening for sleep disorders, a detailed ENT clinical examination including a nasofibroscopy. Each patient then benefits from a sleep recording by ventilatory polygraph.

SUMMARY:
The management of OSA is multidisciplinary. Today, there are many self-evaluation questionnaires aiming at predicting or evaluating the severity of OSA. However, no clinical score takes into account the specificities of the ENT clinical examination, which is a major actor in the management of the disease. The aim of this study is to create a clinical score predictive of the diagnosis and severity of OSA, using already published data, completed with the specificities of the ENT clinical examination.

DETAILED DESCRIPTION:
Obstructive sleep apnea-hypopnea syndrome (OSAHS) is defined as an alteration in nocturnal ventilation related to partial or complete collapse of the upper aerodigestive tract (UAD). The pharyngeal collapse responsible for nocturnal respiratory abnormalities is explained by three factors: anatomical narrowing of the upper airway, increased pharyngeal compliance and loss of efficiency of the pharyngeal dilator muscles. The prevalence of OSA has been estimated to be between 9% and 38%. However, OSA remains under-diagnosed. This syndrome leads, in the absence of treatment, to an overall excess mortality, particularly cardiovascular, and to numerous cardio-metabolic, neurological, psycho-social and road accident complications. Therefore, the identification of patients at risk of OSA through early and targeted screening becomes a public health issue in order to implement an effective treatment to reduce these complications.

VADS examination coupled with nasofibroscopy is a routine examination in ENT consultation. This examination can help to identify patients at risk of OSA and allow its pre-therapeutic evaluation, in order to define the patient's profile and personalize its management. The sites of VADS collapse are multiple. A systematic review on drug induced sleep endoscopy (DISE) found a distribution of obstructive sites of 58.8% for the soft palate, 43.2% for the base of the tongue, 29.9% for the lateral walls of the pharynx and 22.4% for the epiglottis. However, the laryngeal stage also plays a major role in the mechanism of OSA. Endoscopy under induced or natural sleep is a reliable method to identify obstructive sites. However, these techniques require important means (access to the operating room, dedicated hospital room), time, specific equipment and qualified personnel.

The standardized ENT clinical examination coupled with nasofibroscopy is inexpensive, rapid and easily accessible. It allows to identify patients at risk of OSA, to specify the obstructive sites in the VADS and to optimize the therapeutic management by differentiating the patients' profiles.

The objective of this study was to identify anatomical factors predictive of moderate/severe OSA on routine ENT examination in awake patients.

ELIGIBILITY:
Inclusion criteria :

- Adult subjects (> 18 years old), referred to the ENT consultation of the Nancy University Hospital for ENT assessment in the context of OSA or suspicion of OSA, or consultation for the reason "snoring", or presenting clinical signs making OSA suspect.

Non-inclusion criteria:

* Patients suspected of having another sleep disorder (indication for polysomnography)
* Patients with history of upper airway surgery or an ENT tumor

Exclusion criteria:

- Patients with poor quality video recording of nasofibroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included correspond to the patients referred to the ENT consultation at the Nancy University Hospital for clinical screening of sleep apnea/hypopnea syndrome.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
clinical sign and apnea/hypopnea index | Statistical analyses are performed at the end of the recruitment period, when each patient has undergone a clinical examination and a ventilatory polygraph. Measurement date: October 2022.
  Measurement of the association between clinical signs assessed during the ENT examination and the sleep apnea hypopnea index

CONTACTS AND LOCATIONS:
Overall Officials: NGUYEN Duc Trung, PhD, M.P.H, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- LENAY Nicolas, Nancy, France